CLINICAL TRIAL: NCT07338396
Title: A Clinical Study on the Patterns of Traditional Chinese Medicine Syndromes and Efficacy Differences in Lung Cancer Patients Treated With EGFR-TKI
Brief Title: A Prospective Multicenter Study of the Association Between TCM Syndromes and EGFR-TKI Efficacy in Lung Cancer Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Collaborators: Beijing Chest Hospital (Other); Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other); Sichuan Cancer Hospital and Research Institute (Other); Yueyang Hospital of Integrated Traditional Chinese and Western Medicine (Unknown); Affiliated Hospital of Xinxiang Medical University, Henan province (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2025ZD0544601
Record Dates: First submitted 2025-12-16; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Non Small Cell Lung Cancer NSCLC
Keywords: Non Small Cell Lung Cancer NSCLC; Traditional Chinese Medicine Syndromes; Efficacy; EGFR-TKI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Peripheral blood plasma; Peripheral Blood Mononuclear Cells (PBMCs); Fecal specimens; Tongue coating specimens
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Advanced Cohort: Participants in this cohort are patients with stage IIIb-IV non-small cell lung cancer (NSCLC) harboring an EGFR sensitizing mutation, who are receiving or are planned to receive first-line EGFR-TKI therapy within 2 weeks as their first-line treatment.
  Interventions: Drug: EGFR-TKI
- Postoperative Cohort: Participants in this cohort are patients who have undergone complete surgical resection (R0) for NSCLC with an EGFR sensitizing mutation and who are receiving or are planned to receive adjuvant EGFR-TKI therapy within 2 weeks as their postoperative treatment.
  Interventions: Drug: EGFR-TKI

INTERVENTIONS:
Drug: EGFR-TKI — Standard treatment with EGFR tyrosine kinase inhibitors (e.g., gefitinib, erlotinib, osimertinib) for NSCLC. The study observes its association with TCM syndrome patterns.

SUMMARY:
The goal of this observational study is to learn about the relationship between TCM body constitution patterns (called "syndromes") and the effectiveness of EGFR-TKI targeted drugs in patients with lung cancer. Approximately 3000 patients with EGFR-mutant non-small cell lung cancer who are about to start or are already taking EGFR-TKI drugs as part of their regular medical care will be invited to join. Participants will be followed for up to 5 years. During routine clinic visits, researchers will collect their TCM information (such as tongue images and pulse readings) and store small samples of their blood, stool, and tongue coating for future research.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically or histologically confirmed non-small cell lung cancer (NSCLC)
* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Presence of epidermal growth factor receptor (EGFR) mutation confirmed by genetic testing

Postoperative Cohort (must meet all of the above and the following):

* Have undergone curative surgery for lung cancer with R0 resection
* Are planned to receive or are currently receiving postoperative EGFR-TKI adjuvant therapy within 2 weeks

Advanced Cohort (must meet all of the above and the following):

* Meet stage IIIB-IV criteria according to the 9th edition of the American Joint Committee on Cancer (AJCC), or have stage IIIB or below disease but have refused or are unable to tolerate surgical treatment
* Have at least one measurable lesion
* Are planned to receive or are currently receiving first-line EGFR-TKI therapy within 2 weeks

Exclusion Criteria:

* Unable to comply with baseline assessments
* Pregnant or breastfeeding women
* Presence of other uncontrolled malignancies
* Presence of severe brain diseases or psychiatric disorders that affect the patient's ability to communicate or provide informed consent
* Individuals without legal capacity, or those with medical or ethical reasons preventing continued participation in the study
* Refusal to sign the informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll approximately 3000 adult patients with EGFR-mutant non-small cell lung cancer (NSCLC) who are initiating standard EGFR-TKI therapy.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-07 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years.
  Progress free survival defined as the time from first dose of study treatment until the first date of either objective disease progression or death due to any cause.
Disease-Free Survival | From the date of surgery until the date of first documented tumor recurrence, distant metastasis, or death from any cause, assessed up to 5 years.
  From the date of surgery until the date of first documented tumor recurrence, distant metastasis, or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Objective Response Rate | Through study completion, an average of 3 years.
  Objective response rate is defined as the proportion of patients achieving complete (CR) or partial (PR) response according to RECIST V.1.1 criteria.
Disease Control Rate | Through study completion, an average of 3 years.
  Disease control rate is determined by the percentage of patients who achieve CR, PR, or SD as defined by RECIST V.1.1 criteria. This encompasses all instances of CR, PR, and SD (CR + PR + SD).
Overall Survival | From the date of randomization until the date of death from any cause, assessed up to 5 years.
  Overall survival is defined as the time until death due to any cause.
Quality of life evaluation | At the baseline, every 3 months until disease recurrence/progression or the end of the study, assessed up to 3 years.
  According to the requirements of European Organisation for Research and Treatment of Cancer-quality of life core questionnaire (EORTC QLQ-C30)/Lung cancer 29 items (LC 29), the scoring results of each field of the scale were recorded in CRF. The score of this questionnaire ranges between 1 and 4. The higher score indicates the worse quality of life.
Traditional Chinese Medicine Symptom Assessment | At the baseline, every 3 months until disease recurrence/progression or the end of the study, assessed up to 3 years.
  According to the requirements of the MDASI-TCM scale, the scores of each domain were recorded in the CRF. Each item is rated on a numeric scale ranging from 0 to 10, with higher scores indicating greater symptom severity or symptom interference.

OTHER OUTCOMES:
Traditional Chinese Medicine (TCM) Syndrome Classification | At the baseline, every 3 months until disease recurrence/progression or the end of the study, assessed up to 3 years.
  Tongue and pulse characteristics will be collected using standardized and validated tongue diagnosis and pulse diagnosis devices. Standardized symptom information (e.g., fatigue, poor appetite) will be collected by licensed TCM practitioners. Symptoms will be recorded as present or absent without severity grading. Based on tongue, pulse, and symptom information, TCM practitioners will determine and classify each participant's TCM syndrome pattern (e.g., cold syndrome, heat syndrome) at each assessment time point.

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Beijing chest Hospital, Beijing, Beijing Municipality
  - Guang'anmen Hospital of china Academy of chinese Medical Sciences, Beijing, Beijing Municipality
  - Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong
  - Affiliated Hospital of Xinxiang Medical University, Henan province, Weihui, Henan
  - Yueyang Hospital of Integrated Traditional Chinese and Western Medicine, Shanghai, Shanghai Municipality
  - Sichuan Cancer Hospital and Research Institute, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: Undecided